CLINICAL TRIAL: NCT00080145
Title: Risperidone and Behavioral Therapy in Treatment of Children and Adolescents With Autistic Disorder
Brief Title: RUPP PI PDD: Drug and Behavioral Therapy for Children With Pervasive Developmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Denis Sukhodolsky, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U10MH066764 (NIH); U10MH066764 (NIH); U10MH066766 (NIH); U10MH066768 (NIH); DDTR BD-DD
Record Dates: First submitted 2004-03-24; First posted 2004-03-25 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Autistic Disorder; Asperger Syndrome
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder; Asperger Syndrome | interventions — Risperidone; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- risperidone plus parent management training (Active Comparator)
  Interventions: Drug: Risperidone; Behavioral: Behavior Therapy
- risperidone only (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone
Behavioral: Behavior Therapy
  Arms: risperidone plus parent management training

SUMMARY:
This 24-week study will compare the safety and effectiveness of medication treatment alone (risperidone or aripiprazole) to medication treatment in combination with a parent management training program.

DETAILED DESCRIPTION:
PDD can be a profoundly disabling condition across social, emotional, and academic domains. Safe and effective treatments for PDD are needed.

Participants are randomly assigned to receive either risperidone plus parent management training or risperidone alone for 24 weeks. Participants who show deterioration at Week 4 will be offered an alternative mediation treatment, aripiprazole. These participants will remain in their original treatment group (either med alone or med plus parent management training). After 6 months of treatment (Week 24), participants who respond to their treatment will be gradually discontinued from their medication treatment to learn if the response can be sustained without continued medication treatment (This phase of the study was ended in Nov. 2006) Adaptive and behavioral outcomes are assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Autistic Disorder, Asperger's Disorder, or Pervasive Developmental Disorder not otherwise specified
* Weight > 30 lbs
* IQ >= 35 or mental age of at least 18 months

Exclusion Criteria:

* Psychotic Disorder
* History of intolerance or nonresponse to risperidone
* Pregnancy
* History of neuroleptic malignant syndrome

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2004-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Home Situations Questionnaire | Week 24
Vineland Daily Living Skills Scale | Week 24

SECONDARY OUTCOMES:
Irritability subscale-Aberrant Behavioral Checklist | Week 24
Clinical Global Impressions-Improvement (CGI-I) | Week 24

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] McCracken JT, McGough J, Shah B, Cronin P, Hong D, Aman MG, Arnold LE, Lindsay R, Nash P, Hollway J, McDougle CJ, Posey D, Swiezy N, Kohn A, Scahill L, Martin A, Koenig K, Volkmar F, Carroll D, Lancor A, Tierney E, Ghuman J, Gonzalez NM, Grados M, Vitiello B, Ritz L, Davies M, Robinson J, McMahon D; Research Units on Pediatric Psychopharmacology Autism Network. Risperidone in children with autism and serious behavioral problems. N Engl J Med. 2002 Aug 1;347(5):314-21. doi: 10.1056/NEJMoa013171. PMID 12151468
- [Background] Scahill L, McCracken J, McDougle CJ, Aman M, Arnold LE, Tierney E, Cronin P, Davies M, Ghuman J, Gonzalez N, Koenig K, Lindsay R, Martin A, McGough J, Posey DJ, Swiezy N, Volkmar F, Ritz L, Vitiello B. Methodological issues in designing a multisite trial of risperidone in children and adolescents with autism. J Child Adolesc Psychopharmacol. 2001 Winter;11(4):377-88. doi: 10.1089/104454601317261555. PMID 11838820
- [Background] McDougle CJ, Scahill L, McCracken JT, Aman MG, Tierney E, Arnold LE, Freeman BJ, Martin A, McGough JJ, Cronin P, Posey DJ, Riddle MA, Ritz L, Swiezy NB, Vitiello B, Volkmar FR, Votolato NA, Walson P. Research Units on Pediatric Psychopharmacology (RUPP) Autism Network. Background and rationale for an initial controlled study of risperidone. Child Adolesc Psychiatr Clin N Am. 2000 Jan;9(1):201-24. PMID 10674197
- [Derived] Scahill L, Jeon S, Boorin SJ, McDougle CJ, Aman MG, Dziura J, McCracken JT, Caprio S, Arnold LE, Nicol G, Deng Y, Challa SA, Vitiello B. Weight Gain and Metabolic Consequences of Risperidone in Young Children With Autism Spectrum Disorder. J Am Acad Child Adolesc Psychiatry. 2016 May;55(5):415-23. doi: 10.1016/j.jaac.2016.02.016. Epub 2016 Mar 7. PMID 27126856
- [Derived] Calarge CA, Ziegler EE, Del Castillo N, Aman M, McDougle CJ, Scahill L, McCracken JT, Arnold LE. Iron homeostasis during risperidone treatment in children and adolescents. J Clin Psychiatry. 2015 Nov;76(11):1500-5. doi: 10.4088/JCP.14m09258. PMID 26301448
- [Derived] Scahill L, McDougle CJ, Aman MG, Johnson C, Handen B, Bearss K, Dziura J, Butter E, Swiezy NG, Arnold LE, Stigler KA, Sukhodolsky DD, Lecavalier L, Pozdol SL, Nikolov R, Hollway JA, Korzekwa P, Gavaletz A, Kohn AE, Koenig K, Grinnon S, Mulick JA, Yu S, Vitiello B; Research Units on Pediatric Psychopharmacology Autism Network. Effects of risperidone and parent training on adaptive functioning in children with pervasive developmental disorders and serious behavioral problems. J Am Acad Child Adolesc Psychiatry. 2012 Feb;51(2):136-46. doi: 10.1016/j.jaac.2011.11.010. Epub 2011 Dec 23. PMID 22265360
- [Derived] Farmer C, Lecavalier L, Yu S, Eugene Arnold L, McDougle CJ, Scahill L, Handen B, Johnson CR, Stigler KA, Bearss K, Swiezy NB, Aman MG. Predictors and moderators of parent training efficacy in a sample of children with autism spectrum disorders and serious behavioral problems. J Autism Dev Disord. 2012 Jun;42(6):1037-44. doi: 10.1007/s10803-011-1338-2. PMID 21822762
- [Derived] Aman MG, McDougle CJ, Scahill L, Handen B, Arnold LE, Johnson C, Stigler KA, Bearss K, Butter E, Swiezy NB, Sukhodolsky DD, Ramadan Y, Pozdol SL, Nikolov R, Lecavalier L, Kohn AE, Koenig K, Hollway JA, Korzekwa P, Gavaletz A, Mulick JA, Hall KL, Dziura J, Ritz L, Trollinger S, Yu S, Vitiello B, Wagner A; Research Units on Pediatric Psychopharmacology Autism Network. Medication and parent training in children with pervasive developmental disorders and serious behavior problems: results from a randomized clinical trial. J Am Acad Child Adolesc Psychiatry. 2009 Dec;48(12):1143-54. doi: 10.1097/CHI.0b013e3181bfd669. PMID 19858761